CLINICAL TRIAL: NCT06241716
Title: Ultrasound-assisted Versus Real-time Ultrasound-guided Combined Spinal-epidural Anesthesia Via a Paramedian Approach in Elderly Patients: a Randomized Controlled Study
Brief Title: Ultrasound-assisted Versus Real-time Ultrasound-guided Combined Spinal-epidural Anesthesia in Elderly Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Tianzhu Liu, Principal Investigator, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 102114
Record Dates: First submitted 2024-01-04; First posted 2024-02-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-assisted localization, US-AS (Active Comparator)
  Interventions: Procedure: Ultrasound-assisted localization, US-AS; Procedure: Real-time ultrasound guidance, US-RTG
- Real-time ultrasound guidance, US-RTG (Experimental)
  Interventions: Procedure: Ultrasound-assisted localization, US-AS; Procedure: Real-time ultrasound guidance, US-RTG

INTERVENTIONS:
Procedure: Ultrasound-assisted localization, US-AS — In the US-AS group, ultrasonic prescan to determine the best intervertebral space, best puncture Angle and best puncture depth. The optimal puncture section considered by the operator was selected to record the best gap, puncture Angle and depth.
Procedure: Real-time ultrasound guidance, US-RTG — In the US-RTG group, the optimal puncture section considered by the operator was selected and recorded directly in the plane of the paracentral transverse section, out of the plane of the paracentral sagittal section or in the plane of the paracentral sagittal section for real-time ultrasound guided lumbar epidural anesthesia.

SUMMARY:
This study aims to compare the clinical effects of ultrasound-assisted localization and real-time ultrasound-guided combined spinal-epidural anesthesia via paramedian approach in elderly patients

DETAILED DESCRIPTION:
This study aims to compare the clinical effects of ultrasound-assisted localization and real-time ultrasound-guided combined spinal-epidural anesthesia via paramedian approach in elderly patients

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients (≥ 60 years old);
* ASA Grade I to III.

Exclusion Criteria:

* Severe obesity (BMI>35kg/m2);
* Spinal deformity or surgical history;
* Allergic to local anesthetics;
* There are coagulation disorders;
* Communication barriers

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-10-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
First puncture success rate | 1 year
  The proportion of the first successful puncture to the total successful puncture

SECONDARY OUTCOMES:
Procedure time | 1 year
  The time from the contact of the ultrasonic probe to the end of the operation (In seconds).
Positioning time | 1 year
  The time required for pre-scanning and positioning (In seconds).
Depth and width of posterior dural complex | 1 year
  Obtained by ultrasonic measurement (In centimetres).
Skin puncture times | 1 year
  Count the number of skin piercings (In seconds).
Number of redirects | 1 year
  Count the number of needle redirection
Patient satisfaction score (How satisfied the patient is with the whole procedure) | 1 year
  1 is very dissatisfied; 2 is not satisfied; 3 is generally satisfied; 4 are relatively satisfied; A score of 5 is very satisfactory
Operator satisfaction score (How satisfied the patient is with the whole procedure) | 1 year
  1 is very dissatisfied; 2 is not satisfied; 3 is generally satisfied; 4 are relatively satisfied; A score of 5 is very satisfactory

CONTACTS AND LOCATIONS:
Locations (1):
- Tianzhu Liu, Wuhan, Hubei, China

DOCUMENTS (3):
  • Study Protocol (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT06241716/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT06241716/SAP_001.pdf
  • Informed Consent Form (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT06241716/ICF_002.pdf